CLINICAL TRIAL: NCT03022110
Title: Endoscopic Ultrasound-guided Drainage of Pancreatic Pseudocysts: A Multi-center Randomized Controlled Trial
Brief Title: Endoscopic Ultrasound-guided Drainage of Pancreatic Pseudocysts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yiqi Du (Other)
Responsible Party: Sponsor-Investigator, Yiqi Du, Professor, Changhai Hospital
Organization: Changhai Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017010301
Record Dates: First submitted 2017-01-11; First posted 2017-01-16 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Pancreatic Pseudocyst
MeSH Terms: conditions — Pancreatic Pseudocyst

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- plastic stent (Active Comparator): Endoscopic Ultrasound-guided Drainage with plastic stent
  Interventions: Device: Endoscopic Ultrasound-guided Drainage
- lumen-apposing metal stent (LAMS) (Experimental): Endoscopic Ultrasound-guided Drainage with lumen-apposing metal stent
  Interventions: Device: Endoscopic Ultrasound-guided Drainage

INTERVENTIONS:
Device: Endoscopic Ultrasound-guided Drainage — Pancratic pseudocyst drainaged under the guide of Endoscopic Ultrasound

SUMMARY:
The purpose of this study is to compare the effect of lumen-apposing metal stent (LAMS) and traditional plastic stent on the drainage of pancreatic pseudocyst, mainly to observe the cyst recurrence rate of 12 months after treatment.

DETAILED DESCRIPTION:
Inclusion criteria

1. Subject with ages from 18-80 years old
2. Subject with pancreatic pseudocysts confirmed by CT
3. Subject with a history of MSAP or SAP, the pseudocysts were formed more than 3 months
4. The size of pseudocyst is more than 6 cm, and the cyst adjacent to the gastric wall
5. Subject has the symptoms related with the pseudocyst
6. The consent form has been signed

Exclusion criteria

1. Subject is younger than 18 years or older than 80 years
2. Pancreatic pseudocyst communicate with the main pancreatic duct
3. Subject can't accept the endoscopic procedure
4. Pancreatic pseudocyst with infection or subject diagnosed with pancreatic abscess
5. The distance between gastric and the wall of the pseudocyst is more than 1 cm
6. Subject with 2 or more than 2 cysts
7. Subject has blood coagulation dysfunction
8. Pregnant or subject has mental disorders

ELIGIBILITY:
Inclusion Criteria:

1. Subject with ages from 18-80 years old
2. Subject with pancreatic pseudocysts confirmed by CT
3. Subject with a history of MSAP or SAP, the pseudocysts were formed more than 3 months
4. The size of pseudocyst is more than 6 cm, and the cyst adjacent to the gastric wall
5. Subject has the symptoms related with the pseudocyst
6. The consent form has been signed

Exclusion Criteria:

1. Subject is younger than 18 years or older than 80 years
2. Pancreatic pseudocyst communicate with the main pancreatic duct
3. Subject can't accept the endoscopic procedure
4. Pancreatic pseudocyst with infection or subject diagnosed with pancreatic abscess
5. The distance between gastric and the wall of the pseudocyst is more than 1 cm
6. Subject with 2 or more than 2 cysts
7. Subject has blood coagulation dysfunction
8. Pregnant or subject has mental disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2017-02; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Cyst recurrence rate | up to 12 months

SECONDARY OUTCOMES:
Technical success rate | up to 48 hours
Clinical success rate | up to 12 months
Complication rate | up to 12 months

IPD SHARING:
Plan to Share IPD: No